CLINICAL TRIAL: NCT00154375
Title: Phase III Study of Imatinib Mesylate in Combination With Hydroxyurea Versus Hydroxyurea Alone as an Oral Therapy in Patients With Temozolomide Resistant Progressive Glioblastoma
Brief Title: Study of Imatinib Mesylate in Combination With Hydroxyurea Versus Hydroxyurea Alone as an Oral Therapy in Patients With Temozolomide Resistant Progressive Glioblastoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571BDE40
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Results first posted 2011-02-02 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2011-04

CONDITIONS: Glioblastoma Multiforme; Astrocytoma
Keywords: Open label; Imatinib mesylate; hydroxyurea; temozolomide; resistant; protein tyrosine kinases; adenocarcinoma; glioblastoma multiforme; astrocytoma; brain tumor; brain cancer
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Adenocarcinoma; Brain Neoplasms | interventions — Imatinib Mesylate; Hydroxyurea

ARMS (2):
- Imatinib mesylate + hydroxyurea (HU) (Experimental): Imatinib was supplied as 100 mg and 400 mg tablets. Patients in the combination arm were instructed to take a daily oral imatinib dose of 600 mg (600 mg at lunch time) and a daily oral hydroxyurea (HU) dose of 1000 mg (500 mg twice daily; in the morning and at bed time). Every 6 weeks after randomization based on assessment of therapeutic response, either patients continued with above mentioned dosing regimen or switched to receive a daily dose of 800 mg imatinib with 1000 mg HU. Patients were instructed to split the intake, taking 400 mg imatinib with 500 mg HU in the morning, then the same in the evening.
  Interventions: Drug: Imatinib mesylate; Drug: Hydroxyurea
- Hydroxyurea alone (Active Comparator): 1500 mg/day of HU given as 500 mg 3 times daily. Every 6 weeks after randomization and based on assessment of therapeutic response, the patients were either switched to combination arm or continued in monotherapy arm of hydroxyurea.
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Drug: Imatinib mesylate — Imatinib was supplied as 100 mg and 400 mg tablets packaged in polyethylene bottles.
  Other Names: Glivec®
  Arms: Imatinib mesylate + hydroxyurea (HU)
Drug: Hydroxyurea
  Other Names: Litalir®

SUMMARY:
This is a Phase III study comparing Imatinib mesylate and hydroxyurea combination therapy with hydroxyurea monotherapy in patients with temozolomide resistant progressive glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to initiation of any study procedure.
* Patients >= 18 years of age.
* Histological confirmed diagnosis of glioblastoma multiforme / astrocytoma World Health Organization (WHO) grade IV by a reference pathologist
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 or 2.
* Adequate hepatic, renal and bone marrow function as defined by the following: total bilirubin < 1.5 x Upper Limit of Normal (ULN), ALT and AST < 2.5 x ULN, creatinine < 1.5 x ULN, absolute neutrophil count > 1.5 x109/L, platelets > 100 x109/L and hemoglobin > 10 g/dL.
* Female patients of childbearing potential with a negative pregnancy test within 7 days of initiation of study drug dosing. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male and female patients of reproductive potential who agree to employ an effective barrier method of birth control throughout the study, and for up to 3 months following discontinuation of study drug.
* Life expectancy of >3 months.
* MRI available every 6 weeks for disease management
* No intercerebral inflammation
* Irradiation therapy 54 to 62 gy finished or less according to national standard
* Chemotherapy at least 1 temozolomide containing regimen finished, no established chemotherapy regiment available and progression under chemotherapy or in between 6 months following the last chemotherapy.
* Leucocytes > 2.500/µl, to be controlled once a week
* Thrombocytes > 80.000/µl, to be controlled once a week
* Ensured compliance
* Patients who had a second or third resection after disease progression cannot be included earlier than 2 weeks following the resection. MRI should be performed not later than 72 h post operation. If patients are to be included later than 4 weeks after the resection, a new baseline MRI must be performed.

Exclusion Criteria:

* Female patients who are pregnant or breast-feeding.
* Patients who have been treated with any investigational agent(s) within 28 days of the first day of administration of study drug.
* Patients with uncontrolled medical disease such as diabetes mellitus, thyroid dysfunction, neuropsychiatric disorders, infection, angina or Grade 3 or 4 cardiac problems as defined by the New York Heart Association Criteria.
* Patients with other malignant disorders.
* Patient with acute or known chronic liver disease (i.e., chronic active hepatitis, cirrhosis).
* Patients who are known to be HIV positive (no specific tests are required for confirmation of eligibility).
* Expected incompliance according to treatment, treatment diary and examination schedule
* Not confirmed histological diagnosis glioblastoma multiforme/astrocytoma WHO grade IV
* Other drugs with potential cytostatic main or side effect
* No or inadequate chemotherapy or irradiation therapy
* Patients without hematological recovery after previous chemotherapy who have been treated with Chemotherapy within 28 days of the first day of administration of study drug.

Other protocol-specific inclusion /exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2004-10; Primary Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Dülmen, Germany

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Imatinib Mesylate + Hydroxyurea (HU) | Hydroxyurea Alone
Started | 120 | 120
Discontinued Study Treatment | 111 | 104
Not Exposed to Study Treatment | 2 (4 randomized patients didn't receive study treatment were excluded from the safety analyses.) | 2
Completed | 7 | 14
Not Completed | 113 | 106
Not completed — Unsatisfactory therapeutic effect | 25 | 26
Not completed — Adverse Event | 18 | 20
Not completed — Withdrawal by Subject | 14 | 10
Not completed — Death | 5 | 13
Not completed — Study drug no longer required | 5 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Abnormal laboratory value(s) | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Suspected progression of disease | 44 | 30

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Imatinib Mesylate + Hydroxyurea (HU) | Hydroxyurea Alone | Total
Number analyzed (Participants) | 120 | 120 | 240
Age Continuous [Mean (Standard Deviation); unit: years] | 52.1 (11.3) | 50.2 (11.4) | 51.2 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 38 | 88
  Male | 70 | 82 | 152

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression Free Survival (PFS) During the Study Duration
Description: PFS was defined as the time from the date of randomization to the date of the first documented progression according to the MacDonald criteria, or death due to any cause. MacDonald criteria are standard criteria in neurooncology. Tumor assessment was made according to the adapted MacDonald criteria based on the combined evaluation of 1) assessment of the MRI scan for measurable, evaluable, and new lesions (made by the independent external expert too), 2) overall assessment of neurological performance (made by the investigator), 3) concomitant steroid use (as reported by the investigator).
Time Frame: 6 months -1 year
Population: The ITT population consists of all randomized patients, analyzed according to their randomized treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Imatinib Mesylate + Hydroxyurea (HU) | Hydroxyurea Alone
Number analyzed (Participants) | 120 | 120
Percentage of Participants
  6 months | 5.3 [1.0 to 9.7] | 6.6 [2.1 to 11.1]
  12 months | 2.1 [0.0 to 5.0] | 2.1 [0.0 to 5.5]

2. Secondary Outcome: Number of Participants With Death, Other Serious or Clinically Significant Adverse Events (AEs) or Related Discontinuations
Description: National Cancer Institute (NCI)/ National Institute of Health (NIH) provides a grading (severity) scale for each AE term. Grade 3 refers to severe AE and Grade 4 refers to life-threatening or disabling AE. According to FDA 21CFR 314.80, a serious adverse event (SAE) is described as any adverse event that leads to death, is life threatening ( NIH criteria Grade 4), causes or prolongs hospitalization, results in a congenital anomaly, or any other important medical event not described above.
Time Frame: 6 months - 1 year
Population: The safety population consisted of randomized patients with at least one dose of randomized medication.
Measure: Number; unit: Participants
Arm/Group | Imatinib Mesylate + Hydroxyurea (HU) | Hydroxyurea Alone
Number analyzed (Participants) | 118 | 118
Participants
  Deaths | 84 | 91
  Death due to disease progression | 76 | 77
  Serious Adverse Events (SAEs) | 64 | 79
  NCI/NIH Grade 3 (severe) or 4 (life threatening) | 54 | 64
  Suspected to be drug-related | 12 | 12
  Leading to dose adjustment or interruption | 6 | 16
  Leading to permanent discontinuation | 9 | 13

ADVERSE EVENTS:
Description: Safety population = patients who were randomized to either Imatinib + Hydroxyurea (combination)[n=118] or to Hydroxyurea alone [n=118]. Every 6 wks, patients on Hydroxyurea alone switched to combination arm depending on response. So, for the safety analysis Hydroxyurea arm is divided into Hydroxyurea alone [n=118] or switch to combination [n=85].
Groups:
- Imatinib Mesylate + Hydroxyurea (HU): Imatinib was supplied as 100 mg and 400 mg tablets. Patients in the combination arm were instructed to take a daily oral imatinib dose of 600 mg (600 mg at lunch time) and a daily oral hydroxyurea (HU) dose of 1000 mg (500 mg twice daily; in the morning and at bed time). Patients receiving a daily dose of 800 mg imatinib with 1000 mg HU were instructed to split the intake, taking 400 mg imatinib with 500 mg HU in the morning, then the same in the evening.
- Period With Hydroxyurea Alone: 1500 mg/day of HU given as 500 mg 3 times daily.
- Period After Switch to Combination: After every 6 weeks from randomization, depending on the assessment of therapeutic effect, patients were switched from Hydroxyurea (1500 mg/day p.o) to combination arm where patients were instructed to take a daily oral imatinib dose of 600 mg (600 mg at lunch time) and a daily oral hydroxyurea (HU) dose of 1000 mg (500 mg twice daily; in the morning and at bed time).
Arm/Group | Imatinib Mesylate + Hydroxyurea (HU) | Period With Hydroxyurea Alone | Period After Switch to Combination
Serious Adverse Events (participants affected / at risk) | 64/118 | 46/118 | 49/85
Other Adverse Events (participants affected / at risk) | 104/118 | 80/118 | 65/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib Mesylate + Hydroxyurea (HU) (N=118) | Period With Hydroxyurea Alone (N=118) | Period After Switch to Combination (N=85)
ANAEMIA (Blood and lymphatic system disorders) | 2 | 0 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 1 | 2 | 5
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3 | 0 | 2
CARDIAC FAILURE (Cardiac disorders) | 1 | 0 | 0
VISUAL ACUITY REDUCED (Eye disorders) | 0 | 0 | 1
VISUAL DISTURBANCE (Eye disorders) | 1 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 0 | 1
DYSPHAGIA (Gastrointestinal disorders) | 1 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 0 | 1 | 0
STOMATITIS (Gastrointestinal disorders) | 2 | 0 | 0
VOMITING (Gastrointestinal disorders) | 1 | 2 | 0
APLASIA (General disorders) | 1 | 0 | 0
ASTHENIA (General disorders) | 0 | 1 | 1
CHEST PAIN (General disorders) | 0 | 0 | 1
DEATH (General disorders) | 1 | 1 | 2
FATIGUE (General disorders) | 0 | 1 | 0
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 7 | 6 | 2
NECROSIS (General disorders) | 0 | 0 | 1
OEDEMA PERIPHERAL (General disorders) | 1 | 0 | 1
PAIN (General disorders) | 1 | 0 | 0
PERFORMANCE STATUS DECREASED (General disorders) | 1 | 1 | 0
PYREXIA (General disorders) | 1 | 1 | 1
SUDDEN DEATH (General disorders) | 0 | 1 | 0
ASPERGILLOSIS (Infections and infestations) | 0 | 1 | 0
BRONCHITIS (Infections and infestations) | 0 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 1 | 0 | 0
HERPES ZOSTER (Infections and infestations) | 0 | 0 | 1
INJECTION SITE ABSCESS (Infections and infestations) | 1 | 0 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0
PNEUMONIA (Infections and infestations) | 9 | 4 | 5
PNEUMONIA PRIMARY ATYPICAL (Infections and infestations) | 0 | 0 | 1
PULMONARY SEPSIS (Infections and infestations) | 0 | 0 | 1
SEPSIS (Infections and infestations) | 0 | 0 | 2
SINUSITIS (Infections and infestations) | 0 | 0 | 1
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 | 1 | 0
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0
VULVITIS (Infections and infestations) | 1 | 0 | 0
BRAIN CONTUSION (Injury, poisoning and procedural complications) | 1 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 3 | 1 | 3
HEAD INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 0 | 1
SUBDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0 | 0
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 0 | 0 | 1
GENERAL PHYSICAL CONDITION ABNORMAL (Investigations) | 1 | 0 | 0
HEPATIC ENZYME INCREASED (Investigations) | 1 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 | 2 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
INTRACRANIAL TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 1
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 0 | 0 | 2
APHASIA (Nervous system disorders) | 4 | 0 | 0
APRAXIA (Nervous system disorders) | 1 | 0 | 0
BALANCE DISORDER (Nervous system disorders) | 0 | 0 | 2
BRAIN OEDEMA (Nervous system disorders) | 1 | 0 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 | 0 | 1
CONVULSION (Nervous system disorders) | 3 | 4 | 4
COORDINATION ABNORMAL (Nervous system disorders) | 0 | 0 | 2
DEMENTIA (Nervous system disorders) | 0 | 1 | 0
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1 | 0
DISTURBANCE IN ATTENTION (Nervous system disorders) | 1 | 0 | 0
DIZZINESS (Nervous system disorders) | 0 | 0 | 1
DYSPHASIA (Nervous system disorders) | 0 | 0 | 1
EPILEPSY (Nervous system disorders) | 5 | 9 | 9
HEADACHE (Nervous system disorders) | 2 | 5 | 3
HEMIPARESIS (Nervous system disorders) | 8 | 5 | 2
HEMIPLEGIA (Nervous system disorders) | 1 | 2 | 0
INTRACRANIAL PRESSURE INCREASED (Nervous system disorders) | 3 | 3 | 4
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0 | 0
NERVOUS SYSTEM DISORDER (Nervous system disorders) | 0 | 0 | 1
PARESIS (Nervous system disorders) | 1 | 1 | 1
PARTIAL SEIZURES (Nervous system disorders) | 1 | 2 | 4
PSYCHOMOTOR SKILLS IMPAIRED (Nervous system disorders) | 0 | 0 | 1
SOMNOLENCE (Nervous system disorders) | 2 | 1 | 0
SPEECH DISORDER (Nervous system disorders) | 1 | 0 | 0
ABNORMAL BEHAVIOUR (Psychiatric disorders) | 0 | 1 | 0
AGITATION (Psychiatric disorders) | 1 | 0 | 0
ANXIETY (Psychiatric disorders) | 1 | 0 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 4 | 0 | 1
HALLUCINATION (Psychiatric disorders) | 0 | 1 | 0
MENTAL DISORDER (Psychiatric disorders) | 1 | 0 | 0
PERSONALITY DISORDER (Psychiatric disorders) | 1 | 0 | 0
INCONTINENCE (Renal and urinary disorders) | 0 | 0 | 2
OLIGURIA (Renal and urinary disorders) | 0 | 0 | 1
RENAL COLIC (Renal and urinary disorders) | 1 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
BRAIN LOBECTOMY (Surgical and medical procedures) | 0 | 1 | 0
CYSTOSTOMY (Surgical and medical procedures) | 0 | 1 | 0
TUMOUR EXCISION (Surgical and medical procedures) | 3 | 0 | 0
CIRCULATORY COLLAPSE (Vascular disorders) | 1 | 0 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 0 | 0
HYPERTENSION (Vascular disorders) | 0 | 1 | 0
THROMBOSIS (Vascular disorders) | 0 | 1 | 1
VENOUS THROMBOSIS (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib Mesylate + Hydroxyurea (HU) (N=118) | Period With Hydroxyurea Alone (N=118) | Period After Switch to Combination (N=85)
ANAEMIA (Blood and lymphatic system disorders) | 13 | 8 | 13
LEUKOPENIA (Blood and lymphatic system disorders) | 16 | 14 | 14
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 24 | 15 | 17
CUSHINGOID (Endocrine disorders) | 6 | 1 | 5
ABDOMINAL PAIN (Gastrointestinal disorders) | 6 | 3 | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 7 | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 11 | 4 | 5
DIARRHOEA (Gastrointestinal disorders) | 11 | 4 | 4
DYSPEPSIA (Gastrointestinal disorders) | 2 | 6 | 2
NAUSEA (Gastrointestinal disorders) | 28 | 17 | 10
VOMITING (Gastrointestinal disorders) | 21 | 13 | 6
ASTHENIA (General disorders) | 11 | 6 | 9
FATIGUE (General disorders) | 34 | 16 | 18
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 10 | 8 | 4
OEDEMA PERIPHERAL (General disorders) | 29 | 12 | 14
PYREXIA (General disorders) | 6 | 1 | 2
FALL (Injury, poisoning and procedural complications) | 4 | 3 | 5
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 6 | 6 | 1
ANOREXIA (Metabolism and nutrition disorders) | 6 | 2 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 14 | 2 | 6
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6 | 3 | 4
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 | 2 | 6
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 13 | 5 | 3
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 6 | 4 | 2
AMNESIA (Nervous system disorders) | 8 | 2 | 4
APHASIA (Nervous system disorders) | 9 | 4 | 5
CONVULSION (Nervous system disorders) | 6 | 2 | 6
COORDINATION ABNORMAL (Nervous system disorders) | 9 | 9 | 6
DIZZINESS (Nervous system disorders) | 16 | 3 | 7
EPILEPSY (Nervous system disorders) | 13 | 3 | 3
HEADACHE (Nervous system disorders) | 26 | 24 | 16
HEMIPARESIS (Nervous system disorders) | 10 | 7 | 7
LETHARGY (Nervous system disorders) | 6 | 5 | 1
SOMNOLENCE (Nervous system disorders) | 7 | 2 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 9 | 4 | 3
DEPRESSION (Psychiatric disorders) | 3 | 2 | 6
INSOMNIA (Psychiatric disorders) | 4 | 1 | 5
SLEEP DISORDER (Psychiatric disorders) | 6 | 4 | 2
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 4
RASH (Skin and subcutaneous tissue disorders) | 8 | 2 | 0
THROMBOSIS (Vascular disorders) | 1 | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.